CLINICAL TRIAL: NCT01826695
Title: Study of the Effectiveness of a Neurodynamic Intervention in Women With Fibromyalgia.
Brief Title: Neurodynamic Intervention in Fibromyalgia
Acronym: FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant professor, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DF0040UG
Record Dates: First submitted 2013-03-29; First posted 2013-04-08 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, neurodynamic, dexterity
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): 35 women are recruited in order to the inclusion criteria for the study. Placebo controlled. They received only standard treatment without neurodynamic intervention. They are diagnosed with Fibromyalgia attending to the Fibromyalgia Association of Granada. The study include subjects who can complete the assessment battery of tests at the beginning and end.
  Interventions: Other: Placebo group
- Neurodynamic technique group (Active Comparator): 35 women are recruited, diagnosed with Fibromyalgia attending to the Fibromyalgia Association of Granada. The study include subjects who can complete the assessment battery of tests at the beginning and at the end.
  Interventions: Other: Neurodynamic technique group

INTERVENTIONS:
Other: Neurodynamic technique group — Neurodynamic techniques are used in order to move most of the nerves between the neck and hand, including the median nerve, radial and ulnar, brachial plexus, spinal nerves and cervical nerve roots.
  The patient is placed supine position. The treatment will be carry out 3 times per week during 8 weeks.
  Other Names: Neurodynamic sliding technique; Nerve mobilization
  Arms: Neurodynamic technique group
Other: Placebo group — Women in this group realized standard treatment in the Fibromyalgia Association without neurodynamic techniques.
  Other Names: Standard treatment.
  Arms: Placebo group

SUMMARY:
Fibromyalgia is a chronic illness characterised by persistent,widespread muscle pain with generalised hyperalgesia and allodynia. It can be accompanied by other concomitant symptoms like fatigue, sleep disturbances, musculoskeletal disorders, distress and psychological disorders. This condition is very prevalent. It has been reported to be about 2-5% of the general global population.

Fibromyalgia have been reported to have neurodynamic disorders. The purpose of this prospective study was to examine the combined effects of soft tissue mobilization and nerve slider neurodynamic technique on pain and pressure sensitivity in women with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia affects women nine times more than men.The pathophysiology of fibromyalgia is being studied nowadays in order to understand the mechanisms implicated in it.

The treatment propose in this study is a neurodynamic intervention. Neurodynamics is the term used to describe the integration of the morphology, biomechanics and physiology of the nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Fibromyalgia attending to the Fibromyalgia Association of Granada.
* Women who can complete the assessment battery of tests at the beginning and at the end of the study
* Female sex.

Exclusion Criteria:

* Male sex.
* Auditive and visual disturbances.
* Cognitive problems.
* Psychiatric pathology.
* Traumatic pathology of the hand.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Nervous assessment | baseline, 8 weeks
  Changes from baseline to postintervention measured with neurodynamic tests This is to test upper extremities. It moves most of the nerves between the neck and hand, including the median nerve, radial and ulnar, brachial plexus, spinal nerves and cervical nerve roots.
  The patient is placed supine position. It is measured with a goniometer.

SECONDARY OUTCOMES:
Manual dexterity | baseline, 8 weeks
  Changes from baseline to postintervention in dexterity. This is assessed using the Purdue Pegboard Test.
  The Purdue pegboard test is a timed physical test used to measure manual dexterity. Test subjects are asked to place small pins into holes in the pegboard using a specific hand and following a specific process.
Grip strength | baseline, 8 weeks
  Changes from baseline to postintervention in grip strength. This is measured using a Jamar dynamometer with a standard protocol allowing three attempts on each side. During each measurement, patients were sitting with their shoulder adducted and elbow flexed to 90°. The maximum value achieved from all six attempts was used in analyses.
  Kg/cm2
Pressure pain measure | baseline, 8 weeks
  Changes in pain pressure threshold from baseline to 8-weeks intervention. This is going to be measured in three points in upper extremities using the pressure algometer. All assessments were made by the same investigator. All the subjects were trained to familiarize the subjects with the pressure algometry procedure before the measures in an anatomical site different from the chosen sites for this study.

OTHER OUTCOMES:
Anxiety and depression | baseline, 8 weeks
  Changes from baseline to postintervention in anxiety and depression in the participants. Participants completed the Hospital Anxiety and Depression Scale in order to assess these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, phD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torres JR, Martos IC, Sanchez IT, Rubio AO, Pelegrina AD, Valenza MC. Results of an Active Neurodynamic Mobilization Program in Patients With Fibromyalgia Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Oct;96(10):1771-8. doi: 10.1016/j.apmr.2015.06.008. Epub 2015 Jul 2. PMID 26143052